CLINICAL TRIAL: NCT05737407
Title: Lung Ultrasound Guided Choice of Best Positive End-Expiratory Pressure in Neonatal Anesthesia: a Randomized, Controlled Trial
Brief Title: Lung Ultrasound Guided Choice of Best Positive End-Expiratory Pressure in Neonatal Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Principal Investigator, Vittore Buzzi Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022ST251
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Oxygen Toxicity; Anesthesia; Adverse Effect
Keywords: Positive End Expiratory Pressure; Newborn; Atelectasis; Oxygen Toxicity; Lung Ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS-guided Peep (Experimental): After induction of anesthesia and intubation, patients will be briefly turned onto their side and LUS will be performed in the posterior areas of the lung; PEEP will be adjusted in increments of 1 cmH20/minute starting from zero while maintaining visual inspection of LUS up to the point where signs of eventual subpleural consolidations and/or multiple B lines are not present anymore.
  FiO2 will be chosen as the minimum necessary to maintain SpO2 of 97-98%.
  Interventions: Other: LUS-guided choice of Peep
- Standard setting of Peep (Active Comparator): After induction, patients will be similarly scanned with LUS on their side but PEEP will be set at 4 cmH2O independently from results of LUS.
  FiO2 will be chosen as the minimum necessary to maintain SpO2 of 97-98%.
  Interventions: Other: Standard choice of Peep

INTERVENTIONS:
Other: LUS-guided choice of Peep — Choice of Peep guided by lung ultrasound to avoid atelectasis
  Arms: LUS-guided Peep
Other: Standard choice of Peep — Choice of Peep according to standard practice
  Arms: Standard setting of Peep

SUMMARY:
The goal of this RCT is to demonstrate that, in neonatal anesthesia, the use of Lung Ultrasound (LUS) to guide choice of best Positive End-Expiratory Pressure (Peep) - the one that efficiently avoids lung atelectasis - leads to better gas exchange in the lung thus can lead to reduction of FiO2 applied to ventilatory setting in order to achieve same peripheral saturations of oxygen (SpO2).

Specific aims of the study are:

1. to determine if LUS-guided PEEP choice in neonatal anesthesia, compared to standard PEEP choice, can lead to reduction of FiO2 applied to the ventilatory setting in order to maintain same SpO2s.
2. to determine if patients treated with LUS-guided PEEP will develop less postoperative pulmonary complications in the first 24 hours.
3. to compare static respiratory system compliance between groups.
4. to determine if there is a significant difference in hemodynamic parameters and amount of fluids infused or need for vasopressors between the two groups.

DETAILED DESCRIPTION:
The investigators plan to perform a single-center randomised, controlled trial, in compliance with the Helsinki Declaration and local regulatory agreements. Patients of age under two months scheduled for general anesthesia due to elective or urgent surgery will be eligible for enrolment. Eligible cases will be treated by only two experienced anesthesiologists (with more than 10-year experience in pediatric field) who underwent a formal LUS training, in order to reduce operator-dependency of the results. Parental consent to the study will be obtained before entering operatory room.

Both groups will be preliminarily scanned with LUS in the posterior areas before induction of anesthesia, upon entrance into the operatory theatre. Posterior areas of the chest will be defined as the area between the posterior axillary line and the spine, not including the scapular area. This will be further categorized into Upper and Lower as divided by an imaginary line passing through the nipples so that 4 posterior areas are identified: Right Upper Zone, Right Lower Zone, Left Upper Zone, Left Lower zone. For every zone, presence of multiple B lines and subpleural consolidations will be noted. The same ultrasound machine will be used for all cases.

In both groups a standard tidal volume of 6 ml/kg and a standard respiratory rate of 30/min will be applied after anesthesia induction and endotracheal intubation.

Patients will be randomised through the Stata software randomizer just before entering operatory room into one of the 2 following groups:

Intervention group: after induction of anesthesia and intubation, patients will be briefly turned onto their side and LUS will be performed in the posterior areas of the lung; PEEP will be adjusted in increments of 1 cmH20/minute starting from zero while maintaining visual inspection of LUS up to the point where signs of eventual subpleural consolidations and/or multiple B lines are not present anymore.

Control group: after induction, patients will be similarly scanned with LUS on their side but PEEP will be set at 4 cmH2O independently from results of LUS.

FiO2 will be chosen as the minimum necessary to maintain SpO2 of 97-98% in both groups.

Demographic and surgical data will be collected for both groups. Intraoperatively patients will be monitored with standard monitoring systems (SpO2, Heart Rate, Blood Pressure, diuresis, temperature), plus NIRS (Near-Infrared-Spectroscopy); these data will be recorded every 5 minutes. Ventilator settings will also be recorded every 5 minutes. Changes in PEEP or FiO2 needed according to clinical data or need for recruitment manoeuvres will be noted with relative time of occurrence. Major intraoperative complications such as desaturation <90%, hypotension < 5th percentile for age, bradycardia<80 bpm, will be noted. Static compliance will be measured after final PEEP is applied and recorded. Postoperatively, occurrence of PPC in the first 24 hours will be recorded.

Blinding: the anesthesiologist in charge of the case won't be blinded to the group as he/she is the person who will perform LUS and set PEEP and FiO2 for the case. After surgery, the personnel in the ward or ICU, will be blinded to the arm of the study and will record postoperative pulmonary complications. Parents of patients will be blinded too.

ELIGIBILITY:
Inclusion Criteria:

* patients born after 33 weeks of gestationand up to the age of 50 post-conceptional weeks undergoing elective or urgent surgery requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* born at less than 33 weeks of gestation
* patients with signs or symptoms of cardiac or lung abnormalities or diseases
* patients with suspected/confirmed immune diseases, known or suspected metabolic or genetic conditions
* no parental consent is obtained

Ages: 33 Weeks to 50 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of FiO2 applied to the ventilatory setting in order to maintain same SpO2s. | During surgery
  Difference between median SpO2/FiO2 ratio in the two groups

SECONDARY OUTCOMES:
Incidence of Postoperative Pulmonary Complications in the first post-operative 24 hours | In the first 24 hours after the intervention/procedure/surgery
  Comparison of incidence of desaturation (arterial oxyhemoglobin saturation measured with pulsoxymetry < 90% measured and requiring oxygen therapy), need for unplanned postoperative invasive or non invasive ventilation, pneumonia between groups.

OTHER OUTCOMES:
Static compliance of the respiratory system between groups | During surgery
  Static respiratory system Compliance Crs ( ratio of Volume Variation ΔVol to Pressure Variation ΔP)
Need for fluids/vasopressors | During surgery
  Need for fluid replacement and/or vasopressors in the intraoperative phase

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Cildren's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No